CLINICAL TRIAL: NCT01608776
Title: Restoring Equilibrium and Wound Stimulation to Promote Healing Of Non-healing DFUs
Brief Title: RESPOND Restoring Equilibrium and Wound Stimulation to Promote Healing Of Non-healing DFUs
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment delays, business re-allocation of resources
Sponsor: Celleration, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-86036
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SOC - Standard of Care (Active Comparator): Wound cleansing and debridement as needed, moist wound healing dressing, and off-loading
  Interventions: Other: SOC - Standard of Care
- SOC + MIST Therapy (Active Comparator): Wound cleansing and debridement as needed, moist wound healing dressing, off-loading, and MIST treatment
  Interventions: Device: MIST Therapy

INTERVENTIONS:
Device: MIST Therapy — The MIST Therapy System is used as a non-contact method of delivering ultrasound to treat chronic wounds.
  Arms: SOC + MIST Therapy
Other: SOC - Standard of Care — Standard of Care includes wound cleansing and debridement as needed, moist wound healing dressings, and offloading
  Arms: SOC - Standard of Care

SUMMARY:
To evaluate the safety and effectiveness of MIST Therapy in conjunction with Standard of Care (SOC) compared to Standard of Care alone in the treatment of diabetic foot ulcers (DFU).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject of any race and at least 18 to 90 years old
* Lower extremity full thickness diabetic foot ulcer of 30-364 days duration
* Subject's wound must be between 2cm² and 20cm² at screening
* Subject's wound must be at or below the malleolus
* Documented ABI is between 0.8 and 1.2 on the study limb or transcutaneous partial pressure oxygen (TcpO2) > 40 mmHG; or a toe pressure > 40 mmHG; or a Doppler waveform consistent with adequate flow in the foot (biphasic or triphasic waveforms) within 30 days of screening.
* Subject or subject's legally authorized representative understands the nature of the procedure(s) and provides written informed consent prior to study enrollment
* Subject is willing and able to comply with all specified care and visit requirements
* Subject and/or caregiver must be willing and able to learn and perform the duties of dressing changes, and demonstrate the ability to do so.

Exclusion Criteria:

* Index ulcer wound has exposed tendons, ligaments, muscle, or bone
* Index ulcer wound presents with clinical signs of acute infection, suspected or known
* Subjects with evidence of osteomyelitis or cellulitis or gangrene in the study limb
* Subjects with active Charcot's foot on the study limb
* Subjects with amputation above a Trans Metatarsal Amputation (TMA) in the affected limb
* Subjects with active malignancy on the study limb except non-melanoma skin cancer
* Subjects with planned vascular surgery, angioplasty or thrombolysis procedures within the study period
* Subjects within 6 weeks post-operatively of a vascular procedure.
* Subject has had prior skin replacement, negative pressure therapy, or ultrasound therapy applied to the index wound in the 14 days prior to screening
* Subjects who have received oral, or IV antibiotic/antimicrobial agents or medications have been used within 2 days (48 hours) of baseline.
* Subjects who have received topical antibiotic/antimicrobial agents or dressings at the index wound site within 2 days (48 hours) of baseline.
* Subjects currently taking steroids of >10mg dosage
* Subject has received growth factor therapy (e.g., autologous platelet-rich plasma gel, becaplermin, bilayered cell therapy, dermal substitute, extracellular matrix) within 14 days of screening date.
* Subject is currently receiving or has received radiation or chemotherapy within 3 months of randomization.
* Subject has one or more medical condition(s), uncontrolled diabetes (HbA1c > 12), renal, hepatic, hematologic, neurologic, or immune disease that in the opinion of the investigator would make the subject an inappropriate study candidate
* Subject allergic to a broad spectrum of primary & secondary dressing materials, including occlusive dressings and the adhesives on such dressings.
* Female subjects that are pregnant or refuse to utilize adequate contraceptive methods and are of childbearing age during the trial.
* Subject is known to be suffering from a disorder or other situation that the subject or investigator feels would interfere with compliance or other study requirements
* Subject is currently enrolled or has been enrolled in the last 30 days in another investigational device or drug trial

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Wound Reduction | 12 weeks post randomization
  Compare between the treatment groups the index wound area percent reduction, calculated as the difference in cm2 of the randomization measurement to the post four weeks of study treatment measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Vickie Driver, DPM, Principal Investigator
Locations (1):
- Georgetown University Hospital, Washington D.C., District of Columbia, United States